CLINICAL TRIAL: NCT03952546
Title: A Prospective, Randomized, Single-blinded, Non-inferiority Study to Evaluate the Safety and Efficacy of the Saline-coupled Bipolar Sealer Compared to the Unipolar Electrocautery in Primary Unilateral Total Knee Arthroplasty
Brief Title: To Evaluate the Safety and Efficacy of the Saline-coupled Bipolar Sealer in Primary Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS16-0236
Record Dates: First submitted 2016-08-11; First posted 2019-05-16 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Surgical Blood Loss
Keywords: Total Knee Arthroplasty; Surgical Blood Loss; Electrocautery; Perioperative Blood Conservation
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Blinding of the principal investigator and operating staff is not possible. However, all attempts will be made to keep this information from the hospital staff caring for the patients in the postoperative period. The patient and the postoperative hospital staff will be blinded to the treatment arm. The OR staff will be trained not to discuss this information with the patient. During the transition of care from the OR to the Post Anesthetic Care Unit (PACU) the treatment arm will not be included in the verbal patient report. The lack of this information is not required to effectively manage the patient in the postoperative period and will not affect patient care. Postoperatively medical care is managed by the hospitalist, medical doctors specializing in the care of hospitalized patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): Saline-coupled bipolar sealer
  Interventions: Device: Saline-coupled Bipolar Sealer
- Control Arm (Active Comparator): Unipolar electrocautery
  Interventions: Device: Unipolar electrocautery

INTERVENTIONS:
Device: Saline-coupled Bipolar Sealer — The Aquamantys® System is a commercially available device used routinely used in the operating room for a wide variety of surgical cases. It allows for temperatures to stay at approximately 100°C, nearly 200°C less than conventional devices, which produces a tissue effect without the charring associated with other methods. The temperature is sufficient to shrink collagen fibers in the walls of blood vessels, effectively sealing the blood vessels, resulting in the reduction in bleeding from both soft tissue and bone. The device can be used to spot coagulate vessels that are actively bleeding or to broadly paint tissue surfaces to prevent bleeding or treat active oozing.
  Other Names: Aquamantys System(TM)
  Arms: Treatment Arm
Device: Unipolar electrocautery — The Coviden ForceTriad™ energy platform is a full-featured electrosurgical system that provides electrosurgical cutting and coagulation, bipolar functionality, and vessel sealing in a single generator.
  Other Names: Covidien ForceTriad(TM)
  Arms: Control Arm

SUMMARY:
The purpose of this study is to investigate whether the saline-coupled bipolar sealer compared to the unipolar electrocautery provides superior hemostasis in patients undergoing primary unilateral total knee arthroplasty. This will be a prospective, randomized, single-blinded, non-inferiority study in patients scheduled for a primary unilateral total knee arthroplasty (TKA) with Dr. Eugene Krauss or Dr. Ayal Segal. The restriction of this study to two surgeons will limit variations in the outcomes being measured due to differences in surgical technique.

DETAILED DESCRIPTION:
Total joint arthroplasty can result in significant blood loss. Minimizing blood loss has led to multiple blood conservation strategies in orthopaedic procedures. The use of unipolar electrocautery or the saline-coupled bipolar sealer are methods used to reduce intraoperative bleeding. Saline-coupled bipolar sealer technology initially demonstrated promising results in the literature when it was reported that this technology had superior efficacy by reducing blood loss and transfusion requirements in orthopaedic surgery. However, the saline-coupled bipolar sealer technology comes at a significantly higher cost when compared to the unipolar electrocautery. A bipolar electrode costs an additional $450.00 per case, whereas, the unipolar electrocautery catheter is included in all the pre-packaged orthopedic surgical trays. The added cost of the saline-coupled bipolar sealer was offset by the potential savings in the reduced need for blood transfusions. A single blood transfusion is estimated to be $750-$1200. This cost includes both the direct cost of the blood and the additional nursing time needed. Recent publications have challenged the superiority of the saline-coupled bipolar sealer in hemostasis. These randomized clinical trials (RCT) have not supported superiority of this method when compared to standard unipolar electrocautery and the continued use of the saline-coupled bipolar sealer has been questioned. The purpose of this study is to investigate whether the saline-coupled bipolar sealer compared to the unipolar electrocautery provides superior hemostasis in patients undergoing primary unilateral total knee arthroplasty. This will be a prospective, randomized, single-blinded, non-inferiority study in patients scheduled for a primary unilateral TKA with Dr. Eugene Krauss or Dr. Ayal Segal. The restriction of this study to two surgeons will limit variations in the outcomes being measured due to differences in surgical technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for primary unilateral total knee arthroplasty with Dr. Krauss or Dr. Segal
2. Preoperative Hemoglobin >11mg/dL
3. Preoperative platelet count of >150,000
4. Age >18
5. Patient is freely able to provide consent
6. American Society of Anesthesiologists (ASA) classification I-III (Appendix J)
7. Patient willing to complete all study related procedures

Exclusion Criteria:

1. Patients allergic to aspirin
2. Patients with an intolerance to aspirin
3. Patients with a contraindication to Apixaban
4. Any patient who is not a candidate for venous thromboembolism (VTE) risk stratification according to the calculated Caprini Risk Assessment Score. This includes, but is not limited to, any patient who cannot be prescribed ASA 81 mg bid or Apixiban 2.5 mg bid for VTE prophylaxis
5. Patients who for any reason are not a candidate for the use of the monopolar electrocautery
6. History of venous thromboembolism (Deep Vein Thrombosis (DVT), Pulmonary Embolism (PE)) within 12 months prior to the date of surgery
7. Mitral valve replacement or aortic valve replacement with additional risk factor for stroke (atrial fibrillation, previous thromboembolism, left ventricular dysfunction, hypercoagulable conditions)
8. Active cancer
9. Inheritied thrombophilia, eg: Factor V Leiden, Protein C and S deficiencies, Antithrombin deficiency, Prothrombin 20210A mutations
10. Acquired thrombophilia, eg: Lupus anticoagulant, antiphospholipid antibody syndrome
11. Patients taking clopidogrel (Plavix), ticagrelor(Brilinta), or prasugrel (Effient) or any other antiplatelet medication (except for aspirin 81 mg)
12. Patients unable to get intravenous tranexamic acid (TXA) for any reason
13. Patients requiring anticoagulant treatment prior to surgery
14. History of stroke or trans-ischemic attack
15. Serum creatinine > 2.8 mg/dl
16. History of hepatic failure
17. Any medical condition that in the opinion of the investigator would require special fluid management protocols during or after surgery
18. Allergy to TXA
19. Preoperative hemoglobin < 11
20. Preoperative platelets < 150,000
21. Blood transfusion within 1 month of surgery
22. ASA classification IV or V
23. Patients who are unwilling to undergo blood transfusion, if necessary
24. Evidence of active (systemic or local) infection at time of surgery
25. Patients who have habitual opioid use
26. Patients who have a psychiatric or mental illness which could impair the consent process or ability to complete patient-reported questionnaires
27. Fixed motor deficit affecting functional assessment of the knee
28. Patients unable to have spinal anesthesia
29. Patients receiving erythropoietin therapy for anemia
30. Patients who are unable to stop their daily aspirin, aspirin-like products, and/or non-steroidal anti-inflammatory agents 7 days prior to surgery for any reason
31. Patients with a contraindication for the pneumatic tourniquet applied in the operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Krauss, MD, Principal Investigator — Northwell Health
Locations (1):
- Syosset Hospital, Syosset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spahn DR, Goodnough LT. Alternatives to blood transfusion. Lancet. 2013 May 25;381(9880):1855-65. doi: 10.1016/S0140-6736(13)60808-9. PMID 23706802
- [Background] Plymale MF, Capogna BM, Lovy AJ, Adler ML, Hirsh DM, Kim SJ. Unipolar vs bipolar hemostasis in total knee arthroplasty: a prospective randomized trial. J Arthroplasty. 2012 Jun;27(6):1133-7.e1. doi: 10.1016/j.arth.2011.09.016. Epub 2011 Nov 4. PMID 22054904
- [Background] Dunne JR, Malone D, Tracy JK, Gannon C, Napolitano LM. Perioperative anemia: an independent risk factor for infection, mortality, and resource utilization in surgery. J Surg Res. 2002 Feb;102(2):237-44. doi: 10.1006/jsre.2001.6330. PMID 11796024
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Tobias JD. Strategies for minimizing blood loss in orthopedic surgery. Semin Hematol. 2004 Jan;41(1 Suppl 1):145-56. doi: 10.1053/j.seminhematol.2003.11.025. PMID 14872436
- [Background] Esler CN, Blakeway C, Fiddian NJ. The use of a closed-suction drain in total knee arthroplasty. A prospective, randomised study. J Bone Joint Surg Br. 2003 Mar;85(2):215-7. doi: 10.1302/0301-620x.85b2.13357. PMID 12678355
- [Background] Marulanda GA, Ulrich SD, Seyler TM, Delanois RE, Mont MA. Reductions in blood loss with a bipolar sealer in total hip arthroplasty. Expert Rev Med Devices. 2008 Mar;5(2):125-31. doi: 10.1586/17434440.5.2.125. PMID 18331175
- [Background] Weeden SH, Schmidt RH, Isabell G. Haemostatic efficacy of a bipolar sealing device in minimally invasive total knee arthroplasty. J Bone Joint Surg Br Proceedings 2009; 91-B:45.
- [Background] Morris MJ, Berend KR, Lombardi AV Jr. Hemostasis in anterior supine intermuscular total hip arthroplasty: pilot study comparing standard electrocautery and a bipolar sealer. Surg Technol Int. 2010 Oct;20:352-6. PMID 21082586
- [Background] Morris MJ, Barrett M, Lombardi AV Jr, Tucker TL, Berend KR. Randomized blinded study comparing a bipolar sealer and standard electrocautery in reducing transfusion requirements in anterior supine intermuscular total hip arthroplasty. J Arthroplasty. 2013 Oct;28(9):1614-7. doi: 10.1016/j.arth.2013.01.032. Epub 2013 Mar 16. PMID 23507071
- [Background] Zeh A, Messer J, Davis J, Vasarhelyi A, Wohlrab D. The Aquamantys system--an alternative to reduce blood loss in primary total hip arthroplasty? J Arthroplasty. 2010 Oct;25(7):1072-7. doi: 10.1016/j.arth.2009.10.008. Epub 2010 Jan 22. PMID 20097039
- [Background] Strahovnik A, Fokter SK, Kotnik M. Comparison of drainage techniques on prolonged serous drainage after total hip arthroplasty. J Arthroplasty. 2010 Feb;25(2):244-8. doi: 10.1016/j.arth.2008.08.014. Epub 2008 Dec 4. PMID 19056215
- [Background] Johansson T, Engquist M, Pettersson LG, Lisander B. Blood loss after total hip replacement: a prospective randomized study between wound compression and drainage. J Arthroplasty. 2005 Dec;20(8):967-71. doi: 10.1016/j.arth.2005.02.004. PMID 16376249
- [Background] Yang Y, Zhang LC, Xu F, Li J, Lv YM. Bipolar sealer not superior to standard electrocautery in primary total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2014 Oct 10;9:92. doi: 10.1186/s13018-014-0092-5. PMID 25300445
- [Background] Gibon E, Courpied JP, Hamadouche M. Total joint replacement and blood loss: what is the best equation? Int Orthop. 2013 Apr;37(4):735-9. doi: 10.1007/s00264-013-1801-0. Epub 2013 Feb 6. PMID 23385607
- [Background] Eipe NP, Ponniah M. Perioperative blood loss assessment-how accurate? Indian J Anaesth. 2006;50(1):35-38
- [Background] Barsoum WK, Klika AK, Murray TG, Higuera C, Lee HH, Krebs VE. Prospective randomized evaluation of the need for blood transfusion during primary total hip arthroplasty with use of a bipolar sealer. J Bone Joint Surg Am. 2011 Mar 16;93(6):513-8. doi: 10.2106/JBJS.J.00036. PMID 21411700
- [Background] Kamath AF, Austin DC, Derman PB, Clement RC, Garino JP, Lee GC. Saline-coupled bipolar sealing in simultaneous bilateral total knee arthroplasty. Clin Orthop Surg. 2014 Sep;6(3):298-304. doi: 10.4055/cios.2014.6.3.298. Epub 2014 Aug 5. PMID 25177455
- [Background] Abuzakuk T, Senthil Kumar V, Shenava Y, Bulstrode C, Skinner JA, Cannon SR, Briggs TW. Autotransfusion drains in total knee replacement. Are they alternatives to homologous transfusion? Int Orthop. 2007 Apr;31(2):235-9. doi: 10.1007/s00264-006-0159-y. Epub 2006 Jun 8. PMID 16761149
- [Background] Pfeiffer M, Brautigam H, Draws D, Sigg A. A new bipolar blood sealing system embedded in perioperative strategies vs. a conventional regimen for total knee arthroplasty: results of a matched-pair study. Ger Med Sci. 2005 Dec 13;3:Doc10. PMID 19675727
- [Background] Clement RC, Kamath AF, Derman PB, Garino JP, Lee GC. Bipolar sealing in revision total hip arthroplasty for infection: efficacy and cost analysis. J Arthroplasty. 2012 Aug;27(7):1376-81. doi: 10.1016/j.arth.2011.11.016. Epub 2012 Jan 21. PMID 22266048
- [Background] Diedo N, Moore G, et al. Effectiveness of the bipolar sealer in reducing blood loss in total knee arthroplasty. International Journal of Orthopaedic and Trauma Nursing (2013) 17, 29-37
- [Background] Suarez JC, Slotkin EM, Szubski CR, Barsoum WK, Patel PD. Prospective, Randomized Trial to Evaluate Efficacy of a Bipolar Sealer in Direct Anterior Approach Total Hip Arthroplasty. J Arthroplasty. 2015 Nov;30(11):1953-8. doi: 10.1016/j.arth.2015.05.023. Epub 2015 May 19. PMID 26093486
- [Background] Rosenberg AG. Reducing blood loss in total joint surgery with a saline-coupled bipolar sealing technology. J Arthroplasty. 2007 Jun;22(4 Suppl 1):82-5. doi: 10.1016/j.arth.2007.02.018. PMID 17570284
- [Background] Saltzman BM, Oni JK. A Review of Bipolar Sealer Use in Modern Total Joint Arthroplasty. Ann Orthop Rheumatol. 2014 2(2): 1015
- [Background] Marulanda GA, Krebs VE, Bierbaum BE, Goldberg VM, Ries M, Ulrich SD, Seyler TM, Mont MA. Hemostasis using a bipolar sealer in primary unilateral total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2009 Dec;38(12):E179-83. PMID 20145794
- [Background] Lyons ST, Morrison K, Bernasek TL. Sensory neuropathy associated with cauterization using bipolar radio frequency device in primary TKA. Paper presented at: American Academy of Orthopaedic Surgeons Annual Meeting; March 9-13, 2010; New Orleans, LA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the private office practice of the three surgeons who participated in the clinical trials. The first patient signed consent on May 7, 2019. The last patient was consented on 3/10/2021.
Pre-assignment Details: 47 patients were screen failures due to either the blood work not meeting the study enrollment criteria, an exclusion for spinal anesthesia, or the patient decided not to proceed with enrollment in the study.
Groups:
- Saline-Coupled Bipolar Sealer: Device: Saline-coupled Bipolar Sealer The Aquamantys® System is a commercially available device used routinely used in the operating room for a wide variety of surgical cases. It allows for temperatures to stay at approximately 100°C, nearly 200°C less than conventional devices, which produces a tissue effect without the charring associated with other methods. The temperature is sufficient to shrink collagen fibers in the walls of blood vessels, effectively sealing the blood vessels, resulting in the reduction in bleeding from both soft tissue and bone. The device can be used to spot coagulate vessels that are actively bleeding or to broadly paint tissue surfaces to prevent bleeding or treat active oozing.
  Other Names:
  Aquamantys System(TM)
- Unipolar Electrocautery: Device: Unipolar electrocautery The Coviden ForceTriad™ energy platform is a full-featured electrosurgical system that provides electrosurgical cutting and coagulation, bipolar functionality, and vessel sealing in a single generator.
  Other Names:
  Covidien ForceTriad(TM)
Period: Overall Study
Arm/Group | Saline-Coupled Bipolar Sealer | Unipolar Electrocautery
Started | 82 | 82
Completed | 82 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline-Coupled Bipolar Sealer | Unipolar Electrocautery | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 74
  >=65 years | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.3) | 66.1 (8.9) | 65.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 45 | 99
  Male | 28 | 37 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 82 | 82 | 164

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis
Description: Postoperative day 1 estimated blood loss as calculated by the Gross' Formula
Time Frame: Postoperative day 1
Measure: Mean (95% Confidence Interval); unit: milliliters
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 82 | 82
milliliters | 924 [178 to 1861] | 1062 [218 to 2053]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Non-Inferiority — The test for non-inferiority was carried out by calculating the upper 95% confidence limit (one sided confidence interval) for the difference in estimated blood loss (δ = Unipolar electrocautery system - Saline-coupled bipolar sealer), with the margin of inferiority (δ), set at 200 cc; p = 0.1254, t-test, 1 sided

2. Secondary Outcome: Functional Outcomes
Description: Functional outcomes measured by the 2011 "Knee Society Score". The Functional Activities section consists of 4 sub-sections with a total score ranging from 0-100 points. The higher the numerical value the better the outcome. The sub-sections consist of: (1)Walking and Standing 0-30 points (2)Standard Activities 0-30 points (3)Advanced Activities 0-25 points (4)Discretionary Knee Activities 0-15 points.
Time Frame: 8 weeks
Population: 6 participants in the Treatment Arm-Saline-coupled bipolar sealer and 6 participants in the Control Arm-Unipolar electrocautery did not complete the Knee Society Score Questionnaire, therefore, only 76 patients in each of the arms were included in the statistical analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 76 | 76
score on a scale | 56.45 [51.57 to 61.34] | 61.79 [58.19 to 65.39]
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Wound Infection
Description: Participants were assessed for any wound infection within 90 days of surgery.
Time Frame: 90 days postoperatively
Measure: Number; unit: Number of events
Arm/Group | Saline-Coupled Bipolar Sealer | Unipolar Electrocautery
Number analyzed (Participants) | 82 | 82
Number of events | 1 | 3

ADVERSE EVENTS:
Time Frame: 90 days
Description: This clinical trial is designed to compare two commercially available medical devices commonly used in surgical procedures. The devices were used according to the manufacture's guidelines. The clinical trial assessed patients for any return to OR due to bleeding or a hematoma, delayed wound healing, wound infections, any venous thromboembolism events, and skin burns.
Arm/Group | Saline-Coupled Bipolar Sealer | Unipolar Electrocautery
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 1/82 | 3/82
OTHER ADVERSE EVENTS (reported when occurring in more than 1.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saline-Coupled Bipolar Sealer (N=82) | Unipolar Electrocautery (N=82)
Wound Infection (Infections and infestations) | 1 | 3 — Patients were assessed for 90 days postoperatively for any wound infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03952546/Prot_SAP_000.pdf